CLINICAL TRIAL: NCT04807907
Title: Promoting Infant-Directed Speech in Ghana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STU00213766
Record Dates: First submitted 2021-03-12; First posted 2021-03-19 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Infant Development
Keywords: infant directed speech
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Intervention Model Description: The treatment groups are randomly assigned, as follows:
  * Infant Directed Speech (IDS) Video (Treatment; 50%): The participant will be shown a 3-minute video describing the value of IDS and how the participant can use IDS with their child. The participant will receive an IDS-themed wall calendar.
  * Control (50%): No intervention. The participant will receive a regular wall calendar.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infant Directed Speech (IDS) Video + IDS Calendar (Experimental): The participant will be shown a 3-minute video describing the value of IDS and how the participant can use IDS with their child. The participant will receive an IDS-themed wall calendar.
  Interventions: Behavioral: Infant Directed Speech (IDS) Video + IDS Wall Calendar
- Control (No Intervention): No intervention. The participant will receive a regular wall calendar with an image of Stanford.

INTERVENTIONS:
Behavioral: Infant Directed Speech (IDS) Video + IDS Wall Calendar — IDS Video: The IDS video was developed by the research team. It is a simple animation with a voiceover describing the value of IDS and encouraging the viewer to speak to her babies and to tell family members to do so as well. The video has been translated into Dagbani and English (viewers select the language). They may choose to watch it twice.
  Breastfeeding women are told by the surveyor following the video, "For instance, you could talk to your baby in full sentences when your baby is breastfeeding."
  Wall Calendar: The calendar contains images from the video of parents practicing IDS, and key facts about IDS in bullet points. The 12-month calendar contains an empty star next to each week that the respondent can fill in if they perform IDS at least once a day in that week. The calendar also provides a link to a Facebook page where the respondents can re-watch the video or show it to others (https://www.facebook.com/ghanababytalk/videos).
  Arms: Infant Directed Speech (IDS) Video + IDS Calendar

SUMMARY:
The study is a randomized evaluation of a low-cost intervention that encourages mothers and other caregivers to talk to infants, or to engage in what is known as infant-directed speech (IDS) as a way of promoting language and brain development in Tamale and surrounding areas, Ghana.

DETAILED DESCRIPTION:
While parents universally use "baby talk" to soothe an infant or get her attention, engaging in a second form of infant-directed speech (IDS) - talking to young children with complete, if simplified, sentences and a rich variety of words -- varies by socioeconomic status (SES) within societies and across societies. Preliminary evidence collected from Burkina Faso and Ghana, as well as anecdotal experiences in Kenya and Uganda, are consistent with this: It is less common for parents in sub-Saharan Africa to talk to their infants than it is among parents in the US. Because IDS promotes cognitive development of children, gaps in IDS compound the disadvantages that children in poorer families face.

The most likely explanation for the IDS deficit among the poor is inaccurately low expectations about the pace of child development. A large body of literature in the US has shown that the lower the parents' SES, the lower their expectations about when children will master certain cognitive skills, e.g. speaking in a partial sentence of 3 words or more.

The study is a randomized evaluation of a low-cost intervention that encourages mothers and other caregivers to talk to infants, or to engage in what is known as infant-directed speech (IDS) as a way of promoting language and brain development in Tamale and surrounding areas, Ghana.

Parental beliefs about and practices of IDS will be evaluated through data obtained from a series of questions on these topics at baseline, during a short phone follow-up survey, and at endline. This will mainly be self-reported although we hope to explore the observation of said practices at endline. Results of the treatment arm will be compared to that of the comparison group to determine if the intervention is effective. To assess IDS behavior and child language development at endline, the LENA system (Language ENvironment Analysis) which produces two key measures It produced two key measures: adult word count (language the child hears) and conversational turns (the sounds/words the child produces in conversation with adults/others) will be compared among groups. Conditional on funding, there may be a 2-year follow-up survey (i.e. second endline) to measure children's cognitive development.

ELIGIBILITY:
Inclusion Criteria:

* Adult women who visit government health facilities/outreach posts for antenatal, postnatal, or child welfare clinic visits in Tamale and surrounding areas, Ghana.
* Must be age 18 to 40 years old
* Be either pregnant or mothers of young infants at the time of baseline.
* Must speak English or Dagbani (a language local to Tamale and the surrounding areas)

The endline survey will also include child participants.

Child Inclusion Criteria:

* Must be the biological children (or wards) of the baseline respondents
* Must be age 2-18 months old during the endline period

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — adult women and infants they are the primary caregiver for.
Enrollment: 2800 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Adult word count | 10 hours
  Number of words spoken to child
Number of conversational turns | 10 hours
  Number of back-and-forth alternations between a child and an adult during conversation
Self-reported parental beliefs about the value of IDS (Index) | 10 hours
  Questionnaire about at what age the participant believes parents should begin speaking, singing, telling stories, etc. to their child using regular speech (i.e. real words, full sentences). Answers will be used to construct an index.
Self-reported parental IDS behavior (Index) | 10 hours
  Questionnaire about whether the participant uses infant directed speech, and if so, the frequency of this behavior. Answers will be used to construct an index.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

DOCUMENTS (1):
  • Informed Consent Form (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/07/NCT04807907/ICF_000.pdf